CLINICAL TRIAL: NCT00822926
Title: Subcutaneous Botulinum Toxin for Cutaneous Allodynia - Enriched Responder Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SU-01072009-1499; 15601
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A; Sodium Chloride

ARMS (2):
- Placebo then Botox (Experimental): Injection 1: Saline- Subcutaneous injection of saline into scar tissue Injection 2: Botulinum Toxin Type A- Patients receive a subcutaneous injection of Botulinum Toxin Type A into the scar tissue
  Interventions: Drug: Botulinum Toxin Type A; Drug: Saline
- Botox then Placebo (Experimental): Injection 1: Botulinum Toxin Type A- Patients receive a subcutaneous injection of Botulinum Toxin Type A into the scar tissue Injection 2: Saline- Subcutaneous injection of saline into scar tissue
  Interventions: Drug: Botulinum Toxin Type A; Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Patients receive a subcutaneous injection of Botulinum Toxin Type A into the scar tissue
Drug: Saline — Subcutaneous injection of saline into scar tissue

SUMMARY:
Superficial injection of Botulinum toxin has been advocated for cosmetic purposes but has also been reported to be helpful for some pain conditions. The investigators have observed prolonged profound analgesia following subcutaneous superficial injection of Botulinum Toxin Type A (BTA) in patients with certain types of neuropathic pain. the investigators propose to study if addition of BTA extends pain relief compared to placebo when injected subcutaneously into areas of cutaneous allodynia (the property that a normally non-noxious stimulus is perceived as painful).

DETAILED DESCRIPTION:
Patients with post-herpetic neuralgia, complex regional pain syndrome, and post-surgical neuromatous pain patients have marked cutaneous allodynia. Touching their skin with normally non-painful stimuli results in pain. Injected local anesthetics are often effective in providing temporary relief. In the course of clinical practice the investigators have observed that a number of patients with cutaneous allodynia have had marked persistent benefit from subcutaneous injection of Botulinum toxin Type A.

Rather than killing targeted neurons, Botulinum toxin type A inhibits release of acetylcholine from cholinergic nerve terminals in a prolonged but ultimately reversible manner. Neuropathic pain and its hallmark allodynia are classically difficult to treat. Standard treatment with tricyclic antidepressants, anti-epileptic drugs, opiates and spinal cord stimulation is frequently disappointing leaving patients with refractory pain. Surgical or percutaneous ablation of involved nerves has fallen out of favor among many due to disappointing results.

A pilot study is needed to assess the efficacy of superficially injected Botulinum Toxin type A for treatment of cutaneous allodynia and spontaneous pain among patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain (greater than 2/10) of duration more than 6 months despite previous therapy, excluding botox injection
* The patient exhibits at least 80% pain relief following injection of local anesthetic subcutaneously into scar as assessed by change in NRS
* Patient reports more than 3 weeks of greater than 50% pain relief from previous botox injection
* The patient reports the presence of hyperalgesia, allodynia, dysesthesia, or hypoesthesia surrounding the scar in the absence of the botox injection
* Age 18-100
* Ability to read, write, and converse in English, provide informed consent, and follow study procedures

Exclusion Criteria:

* Any neuromuscular disorder such as myasthenia gravis, eaton lambert, muscular dystrophy
* Any ongoing legal action related to their pain
* Allergy to local anesthetics
* Any ongoing disability claim
* Currently being treated for any severe psychiatric disorder, including anxiety or depression
* History of any adverse reaction to botulinum toxin
* History of botulism
* Untreated infection
* Coagulopathy
* (Females) - positive pregnancy test
* Surgery in the last 6 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Carroll, Principal Investigator — Stanford University; Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: First Injection Visit
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Washout (Varies Based on Scheduling)
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Second Injection Visit
Arm/Group | Placebo Then Botox | Botox Then Placebo
Started | 2 | 3
Completed | 1 | 2
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Botox | Botox Then Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (4.24) | 48.5 (7.78) | 48.75 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Analgesic Failure
Description: Participants completed the Pain Numeric Rating Scale everyday after the injections. Outcome measure represents the number of days before pain returned to baseline levels.
Time Frame: Duration of trial (2-20 months, depending on how long pain relief lasts)
Population: A total of 3 participants completed the study (1 received Placebo first then Botox, 2 received Botox first then Placebo). Each of those 3 participants received both Placebo and Botox, as represented in the overall number of participants analyzed for both treatments.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo: Saline- Subcutaneous injection of saline into scar tissue
- Botox: Botulinum Toxin Type A- Patients receive a subcutaneous injection of Botulinum Toxin Type A into the scar tissue
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 3 | 3
days | 120.67 (166.79) | 20.67 (22.72)

2. Secondary Outcome: Improvement in Psychosocial Function as Assessed by Outcomes as Dictated by the IMMPACT Guidelines
Description: The Beck Depression Inventory was used to assess psychosocial function. Scores were measured at baseline, their final questionnaire following the first injection visit, and their final questionnaire following their second injection visit. Scores range from 0-63, with lower scores representing less severe depression symptoms and higher scores representing more severe depression symptoms.
Time Frame: Duration of trial (2-20 months, depending on how long pain relief lasts)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Baseline | Placebo | Botox
Number analyzed (Participants) | 3 | 3 | 3
Units on a scale | 12.33 (3.79) | 8 (7.21) | 8 (4.36)

3. Secondary Outcome: NRS Score Three Weeks After Injection
Description: Pain scores were measured at baseline, 3 weeks after placebo, and 3 weeks after botox. Scores range from 0 (no pain) to 10 (severe, disabling pain).
Time Frame: 3 weeks after injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Baseline | Placebo | Botox
Number analyzed (Participants) | 3 | 3 | 3
Units on a scale | 3.39 (2.46) | 0.86 (0.7) | 3.2 (2.18)

ADVERSE EVENTS:
Arm/Group | Placebo Then Botox | Botox Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Then Botox (N=2) | Botox Then Placebo (N=3)
Stomach flu (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes